CLINICAL TRIAL: NCT07077668
Title: Extended Study of RAG-17 in the Treatment of Amyotrophic Lateral Sclerosis Patients With SOD1 Gene Mutation
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice-President of Beijing Tiantan Hospital,Chief Scientist of Neurology Center, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-A-2025020
Record Dates: First submitted 2025-06-20; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Amyotrophic lateral sclerosis; RAG-17; SOD1
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Patients who meet the inclusion and exclusion criteria are required to come to the hospital at the following time points to complete the intrathecal bolus injection of quantitative RAG - 17, relevant examinations, and evaluations by the research physicians: baseline, 60 ± 3 days, 120 ± 3 days, 180 ± 3 days, 240 ± 3 days, 300 ± 3 days, 360 ± 3 days, 450 ± 3 days, 540 ± 3 days. An online follow - up will be conducted at 570 ± 3 days.
  Interventions: Drug: A sterile aqueous solution of RAG - 17 preparation (sodium salt)

INTERVENTIONS:
Drug: A sterile aqueous solution of RAG - 17 preparation (sodium salt) — Patients who meet the inclusion and exclusion criteria are required to come to the hospital at the following time points to complete the intrathecal bolus injection of RAG - 17 for 150 mg: baseline, 60 ± 3 days, 120 ± 3 days, 180 ± 3 days, 240 ± 3 days, 300 ± 3 days, 360 ± 3 days, 450 ± 3 days, 540 ± 3 days.

SUMMARY:
This study primarily evaluates the safety, tolerability, and efficacy of RAG - 17 in adult ALS patients with SOD1 - mutated genes in the real - world setting.

DETAILED DESCRIPTION:
Based on the results of the previous investigator - initiated trial (IIT) of RAG - 17 in the treatment of SOD1 - ALS, this study further planned to conduct another small - sample real - world research. By administering regular and quantitative intrathecal injections of RAG - 17 to subjects who meet the inclusion criteria of the study, the safety, tolerability, and efficacy of RAG - 17 in adult ALS patients with SOD1 - mutated genes in the real - world setting will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ Age ≤ 75 years old, regardless of gender.
* ALS patients with confirmed SOD1 gene mutations (known SOD1 mutation sites with reported relevant disease progression).
* The diagnosis meets the criteria for definite or probable familial or sporadic ALS in the El Escorial diagnostic criteria for amyotrophic lateral sclerosis revised by the World Federation of Neurology.
* The patient himself/herself or their legal representative clearly understands, voluntarily participates in this study, and signs the informed consent form.

Exclusion Criteria:

* Patients with SOD1 mutation sites occurring at nucleotides 44 - 66 (counting from the start of SOD1 protein translation) and patients with P.F21C mutation.
* Patients diagnosed with other mental illnesses according to the DSM - V diagnostic criteria, or those with obvious suicidal intent.
* Patients with severe hepatic insufficiency, severe renal insufficiency, or severe cardiac insufficiency. (Severe hepatic insufficiency refers to an ALT value ≥ 2.0 times the upper limit of normal or an AST value ≥ 2.0 times the upper limit of normal; severe renal insufficiency refers to a CRE ≥ 1.5 times the upper limit of normal or an eGFR < 40 mL/min/1.73m²; severe cardiac insufficiency refers to a NYHA score of 3 - 4.)
* Patients with a history of alcohol or drug abuse.
* Pregnant, lactating patients, those with a possibility of pregnancy, or patients planning to become pregnant.
* Patients who have received any vaccination within 28 days.
* Patients who are unable to cooperate with the follow - up for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | Baseline to 570 days
  Incidence of adverse events and serious adverse events within 570 days after treating SOD1 - ALS patients with RAG - 17 in the real world, and number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) V5.0.
ALSFRS-R score | baseline, 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, 540±3 days, and 570±3 days
  Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score (ALSFRS-R scores from 0 to 48, score decline indicates worse outcome of ALS patients, or disease progression and disability)

SECONDARY OUTCOMES:
The level of SOD1 protein in cerebrospinal fluid | baseline, 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, and 540±3 days
  The level of SOD1 protein in the cerebrospinal fluid of ALS patients is positively correlated with the disease severity. Changes in the level of SOD1 protein in cerebrospinal fluid relative to the baseline at 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, and 540±3 days after treating SOD1 - ALS patients with RAG - 17 in the real - world setting
Plasma neurofilament light chain protein (NFL) level | baseline, 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, and 540±3 days
  The level of neurofilament light chain (NFL) in blood of ALS patients. Value increase indicates neuroinflammation or nerve damage. Changes in plasma neurofilament light chain protein (NFL) levels relative to the baseline at 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, and 540±3 days after treating SOD1 - ALS patients with RAG - 17 in the real world
Invasive mechanical ventilation | From date of randomization until the date of first documented event about invasive mechanical ventilation. The assessment period is up to 30 months.
  The time of occurrence of invasive mechanical ventilation after treating SOD1-ALS patients with RAG-17 in the real world
Gastrostomy | From date of randomization until the date of first documented event about gastrostomy. The assessment period is up to 30 months.
  The time of occurrence of gastrostomy after treating SOD1-ALS patients with RAG-17 in the real world
Death | From randomization date to date of death from any cause. The assessment period is up to 60 months.
  The time of occurrence of death after treating SOD1-ALS patients with RAG-17 in the real world
Muscle strength (MRC Scale) | baseline, 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days and 540±3
  Medical Research Council Scale (MRC Scale) is an assessment that is used to measure the change in muscle strength. MRC Scales ranges from grade 0 to grade 5, where grade 0 means no muscle contraction, grade 5 means muscle has full strength. Changes in muscle strength relative to the baseline at 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days and 540±3 days after treating SOD1-ALS patients with RAG-17 in the real world
ALSAQ-40 | baseline，60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, 540±3 days and 570±3 days
  Change in Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) score (from 40 to 200, score decline indicates worse outcome of ALS patients, or disease progression and disability). Changes in ALSAQ-40 relative to the baseline at 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, 540±3 days and 570±3 days after treating SOD1 - ALS patients with RAG - 17 in the real world
EQ-5D-5L | baseline，60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, 540±3 days and 570±3 days
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that is used to measure the changes in the quality of life. EQ-5D-5L contains 5 domains including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each domain is scored on a 5-level severity from Level1(no difficulty) to Level5 (extreme difficulty). Changes in EQ-5D-5L relative to the baseline at 60±3 days, 120±3 days, 180±3 days, 240±3 days, 300±3 days, 360±3 days, 450±3 days, 540±3 days and 570±3 days after treating SOD1 - ALS patients with RAG - 17 in the real world.

CONTACTS AND LOCATIONS:
Overall Officials: Wang YiLong, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No